CLINICAL TRIAL: NCT00695292
Title: Phase II Study of Irinotecan, Carboplatin, and Sunitinib in the First Line Treatment of Extensive-Stage Small Cell Lung Cancer
Brief Title: Irinotecan, Carboplatin, and Sunitinib in First Line Extensive-Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI LUN 156
Record Dates: First submitted 2008-06-09; First posted 2008-06-11 (Estimated); Results first posted 2013-02-15 (Estimated); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Small Cell Lung Cancer
Keywords: Small Cell Lung Cancer; Extensive Stage; irinotecan; carboplatin; sunitinib
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Irinotecan; Carboplatin; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): Patients in the study will receive the following for the duration of the study: irinotecan 60 mg/m2 intravenously on Days 1, 8, and 15 and carboplatin AUC=4 on Day 1. The study will consist of 28-day cycles, to a maximum of 6 cycles of therapy with irinotecan and carboplatin. After treatment with irinotecan and carboplatin, sunitinib will be given alone as maintenance therapy in all patients who have achieved study entry hematologic criteria and who do not have progressive disease or severe toxicity. During sunitinib maintenance therapy, patients will receive sunitinib at 25 mg orally daily. Sunitinib maintenance therapy will continue until progressive disease or irreversible toxicity occurs.
  Re-staging will be performed every 2 cycles (every 8 weeks) during the study.
  Interventions: Drug: irinotecan; Drug: Carboplatin; Drug: sunitinib

INTERVENTIONS:
Drug: irinotecan — irinotecan 60 mg/m2 intravenously (IV) on Days 1, 8, and 15
  Other Names: Camptosar
Drug: Carboplatin — carboplatin AUC=4 on Day 1
  Other Names: Paraplatin
Drug: sunitinib — sunitinib 25 mg orally (PO) daily after initial chemotherapy
  Other Names: Sutent

SUMMARY:
This proposed Phase II trial will investigate the combination of irinotecan and carboplatin followed by sunitinib in the first-line treatment of patients with extensive-stage SCLC.

DETAILED DESCRIPTION:
Irinotecan/platinum regimens are emerging as standard treatments for patients with extensive-stage disease. The irinotecan/carboplatin doses that will be used in this study have been used in two previous Phase II SCLC trials, and were found to be extremely well tolerated (Thompson et al. 2005; Spigel et al. 2007). Adding a novel, minimally toxic agent to this regimen may further enhance efficacy in this patient population without contributing to toxicity. This trial will evaluate the use of sunitinib following 6 cycles of treatment with chemotherapy in the treatment of SCLC.

The trial will be performed under the leadership of SCRI, a community-based, multi-center, clinical trial organization.

ELIGIBILITY:
Inclusion Criteria:

1. Cytologically and/or histologically confirmed small-cell lung cancer with extensive-stage disease.
2. Measurable or evaluable disease.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1.
4. Adequate bone marrow function, as defined by: absolute neutrophil count (ANC) >1,500/µL; platelets >100,000/µL; hemoglobin >=9.0 g/dL.
5. Normal organ function, defined as follows: aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <=2.5 × the upper limit of normal (ULN), or AST and ALT <=5 × the ULN if liver function abnormalities are due to underlying malignancy; total serum bilirubin <=1.5 × the ULN; serum creatinine <=1.5 × the ULN.
6. Resolution of all acute toxic effects of prior therapy or surgical procedures to grade <=1.
7. Women of childbearing potential and men with partners of childbearing potential must agree to use a form of birth control that is acceptable to their physician to prevent pregnancy during treatment.
8. Patients must be informed of the investigational nature of this study and sign an informed consent form.
9. Patients who have treated brain metastases >=4 weeks out (with surgery and/or radiation therapy) and who have no evidence of central nervous system (CNS) progression. Steroid use should be discontinued before study treatment begins.

Exclusion Criteria:

1. Patients who are pregnant or breastfeeding.
2. Patients may not have received other agents (either investigational or marketed) which act by anti-angiogenic mechanisms. Angiogenesis inhibitors include (but are not limited to): thalidomide, sorafenib, bevacizumab.
3. Patients who have had previous chemotherapy or radiation therapy for extensive-stage disease will be excluded. Palliative radiation (e.g., for bone disease) or radiation for cranial metastasis is acceptable if the patient has recovered from any adverse effects.
4. Previous treatment with sunitinib.
5. Myocardial infarction, severe or unstable angina, coronary/peripheral artery bypass graft, congestive heart failure (CHF), cerebrovascular accident (including transient ischemic attack), or pulmonary embolism within 6 months prior to study initiation.
6. Ongoing cardiac dysrhythmias of National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) grade >=2, atrial fibrillation of any grade, or prolongation of the QTc interval to >450 msec (for males) or >470 msec (for females).
7. Uncontrolled hypertension (i.e., blood pressure >150 mm Hg that cannot be controlled with standard anti-hypertensive agents).
8. Active brain metastasis. (Patients who had brain metastases treated with radiation or surgery and have no evidence of progressive brain metastases at least 4 weeks later are eligible).
9. Patients who have had major surgical procedure, open biopsy, or significant traumatic injury with 28 days (4 weeks) of study initiation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2008-06; Primary Completion 2011-06 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R Spigel, M.D., Study Chair — SCRI Development Innovations, LLC
Locations (10):
- United States (10):
  - Florida Cancer Specialists, Fort Myers, Florida
  - Florida Hospital Cancer Insitute, Orlando, Florida
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - St. Louis Cancer Care, Chesterfield, Missouri
  - Oncology Hematology Care, Cincinnati, Ohio
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Chattanooga Oncology Hematology Associates, Chattanooga, Tennessee
  - Tennessee Oncology, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Groups:
- Irinotecan, Carboplatin, Sunitinib: Patients receive irinotecan 60mg/m2 IV on days 1, 8, and 15 and carboplatin AUC=4 on day 1 of each 28-day cycle. After completion of 6 cycles, patients receive only sunitinib 25 mg daily by mouth.
Period: Overall Study
Arm/Group | Irinotecan, Carboplatin, Sunitinib
Started | 37
Completed | 37
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Irinotecan, Carboplatin, Sunitinib
Number analyzed (Participants) | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 21
Region of Enrollment [Number; unit: participants]
  United States | 37

OUTCOME MEASURES:

1. Primary Outcome: One-year Survival, The Percentage of Patients Who Are Alive One Year After Completing Protocol Treatment
Time Frame: 18 months
Population: The original study design administered sunitinib concurrently with irinotecan/carboplatin. After the first three patients enrolled experienced severe myelosuppression, the treatment plan was modified to delay sunitinib until after completion of combination therapy. Only patients treated under the revised plan are included in the results analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Irinotecan, Carboplatin, Sunitinib
Number analyzed (Participants) | 34
percentage of participants | 54

2. Secondary Outcome: Overall Response Rate (ORR), the Percentage of Patients Who Experience an Objective Benefit From Treatment
Description: Objective benefit is defined as substantial (30% or greater) shrinkage in tumor volume per RECIST 1.0.
Time Frame: 18 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Irinotecan, Carboplatin, Sunitinib
Number analyzed (Participants) | 34
percentage of participants | 59 [41 to 75]

3. Secondary Outcome: Time to Progression
Description: Time To Progression (TTP) was defined as the interval between the start date of treatment and the date of occurrence of progressive disease
Time Frame: 18 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Irinotecan, Carboplatin, Sunitinib
Number analyzed (Participants) | 34
months | 7.6 [5.7 to 9]

4. Secondary Outcome: Median Overall Survival
Description: Overall survival was defined as the interval between the date of study entry until the date of death.
Time Frame: 18 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Irinotecan, Carboplatin, Sunitinib
Number analyzed (Participants) | 34
months | NA [NA to NA] — The median overall survival (OS) has not been reached due to insufficient observed events

5. Secondary Outcome: Number of Participants Experiencing Treatment Related Toxicity
Description: The toxicity assessments were made according to the common terminology criteria for adverse events (CTCAE version 3.0) of the National Cancer Institute. Number of participants with Grade 1 to 5 adverse events are reported here.
Time Frame: 18 months
Population: Toxicity was evaluated in all patients who received at least 1 dose of therapy. The original study design administered sunitinib concurrently with irinotecan/carboplatin. After the first three patients enrolled experienced severe myelosuppression, the treatment plan was modified to delay sunitinib until after completion of combination therapy. Only patients treated under the revised plan are included in the results analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Irinotecan, Carboplatin, Sunitinib
Number analyzed (Participants) | 34
Participants | 32

ADVERSE EVENTS:
Groups:
- Intervention: Patients in the study will receive the following for the duration of the study: irinotecan 60 mg/m2 intravenously on Days 1, 8, and 15 and carboplatin AUC=4 on Day 1. The study will consist of 28-day cycles, to a maximum of 6 cycles of therapy with irinotecan and carboplatin. After treatment with irinotecan and carboplatin, sunitinib will be given alone as maintenance therapy in all patients who have achieved study entry hematologic criteria and who do not have progressive disease or severe toxicity. During sunitinib maintenance therapy, patients will receive sunitinib at 25 mg orally daily. Sunitinib maintenance therapy will continue until progressive disease or irreversible toxicity occurs.
Arm/Group | Intervention
Serious Adverse Events (participants affected / at risk) | 18/37
Other Adverse Events (participants affected / at risk) | 34/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=37)
Death (General disorders) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Platelets (Blood and lymphatic system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
ARDS (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Disease Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4)
Infection - Sepsis (Infections and infestations) | 2 (2)
Diverticulitis (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Pain - Chest (Cardiac disorders) | 1 (1)
Intractable Pain (General disorders) | 1 (1)
Infection - Pneumonia (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=37)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (15)
Anorexia (Gastrointestinal disorders) | 11 (21)
AST (Metabolism and nutrition disorders) | 2 (3)
Ataxia (Nervous system disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 13 (40)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (12)
Creatinine (Metabolism and nutrition disorders) | 2 (2)
Dehydration (Gastrointestinal disorders) | 11 (11)
Diarrhea (Gastrointestinal disorders) | 20 (64)
Dizziness (Nervous system disorders) | 7 (16)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 14 (58)
Edema: Limb (Blood and lymphatic system disorders) | 7 (20)
Esophagitis (Gastrointestinal disorders) | 4 (4)
Fatigue (General disorders) | 30 (117)
Febrile Neutropenia (Infections and infestations) | 2 (2)
Fever (General disorders) | 6 (7)
Gait/Walking (Musculoskeletal and connective tissue disorders) | 2 (2)
Heartburn (Gastrointestinal disorders) | 8 (22)
Hemoglobin (Blood and lymphatic system disorders) | 34 (117)
Hemorrhage - Nose (Blood and lymphatic system disorders) | 2 (2)
Hemorrhage, Pulmonary/Upper Respiratory (Blood and lymphatic system disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (12)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2)
Hypertension (Cardiac disorders) | 2 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 5 (9)
Hypokalemia (Metabolism and nutrition disorders) | 8 (12)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (10)
Hyponatremia (Metabolism and nutrition disorders) | 9 (10)
Hypotension (Cardiac disorders) | 6 (15)
Infection - Other (Infections and infestations) | 2 (2)
Infection - Pneumonia (Infections and infestations) | 5 (6)
Insomnia (General disorders) | 8 (12)
Leukocytes (Blood and lymphatic system disorders) | 31 (93)
Mood Alteration - Anxiety (Psychiatric disorders) | 5 (16)
Mucositis/Stomatitis (Gastrointestinal disorders) | 8 (10)
Muscle Weakness (Extremity-Lower) (Musculoskeletal and connective tissue disorders) | 3 (4)
Muscle Weakness (NOS) (Musculoskeletal and connective tissue disorders) | 2 (3)
Nausea (Gastrointestinal disorders) | 27 (72)
Neuropathy: Motor (Nervous system disorders) | 2 (3)
Neuropathy: Sensory (Nervous system disorders) | 4 (9)
Neutrophils (Blood and lymphatic system disorders) | 28 (64)
Pain - Muscle (General disorders) | 4 (5)
Pain - Other (General disorders) | 4 (10)
Pain - Abdomen (General disorders) | 8 (19)
Pain - Back (General disorders) | 7 (17)
Pain - Bone (General disorders) | 4 (7)
Pain - Chest (General disorders) | 8 (12)
Pain - Dental/Teeth/Periodontal (General disorders) | 2 (3)
Pain - Head (General disorders) | 7 (12)
Pain - Joint (General disorders) | 11 (28)
Pain - Limb (General disorders) | 6 (12)
Platelets (Blood and lymphatic system disorders) | 23 (53)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pulmonary, Other (COPD) (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 3 (8)
Renal Failure (Renal and urinary disorders) | 2 (2)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Rigors/Chills (General disorders) | 2 (2)
Superventricular Arrhythmia (Atrial Fibrillation) (Cardiac disorders) | 2 (2)
Supraventricular Arrhythmia (Tachycardia) (Cardiac disorders) | 3 (4)
Sweating (General disorders) | 4 (5)
Taste Alteration (Gastrointestinal disorders) | 5 (9)
Tremor (Nervous system disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 14 (40)
Weight Gain (Metabolism and nutrition disorders) | 2 (3)
Weight Loss (Metabolism and nutrition disorders) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 days but ≤180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites.